CLINICAL TRIAL: NCT02383459
Title: Longitudinal Study of Food Liking in Eatrly Childhood
Brief Title: Observatory of Food Preferences in Infants and Children
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Burgundy (Other)
Responsible Party: Sponsor
Other Study IDs: OPALINE
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
Food habits form early in infancy and are likely to track into childhood until the beginning of adulthood. Understanding the factors driving the acceptance of foods in the early years is therefore of particular importance, since these foods will form the basis of a child's future food repertoire. This is especially important for vegetables, which consumption is recommended at all stages of life but is below the recommended levels and which acceptance is difficult to promote during late childhood.

The objective of the present study was to unravel the respective contribution of maternal feeding practices, of children's rate of exposure to vegetables and of children's sensory reactivity factors over the course of the first two years, to explain the development of liking for vegetables at the age of 2 years. This analysis took advantage of data recorded in a prospective cohort of children recruited before birth and followed up longitudinally until the age of 2 years.

DETAILED DESCRIPTION:
This study is a cohort study with the aim to evaluate prospectively food liking in children, at to relate this outcome to children's food experience, acceptance of taste and olfactory stimulation, and to parental feeding style.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers older than 18 years

Exclusion Criteria:

* Food allergies in the infant, as observed after the infant's birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Food likes (Evaluation of food likes for a list of 257 foods) | 1-year prospective data collection
  Evaluation of food likes for a list of 257 foods